CLINICAL TRIAL: NCT07104422
Title: An Epidemiological and Long-Term Endpoint Registry Study on Disease-Syndrome Correlation Patterns in Comorbid Population With Diabetes and Ischemic Cardio-Cerebrovascular Disease
Acronym: Diabetes
Status: Not yet recruiting | Type: Observational
Sponsor: Guangzhou University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 2023ZD0505601; An Epidemiological and Long-Te (Other Grant/Funding Number: Ministry of Science and Technology)
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Type 2 Diabetes Mellitus (T2DM); Cardiovascular Complications
Keywords: Diabetes comorbidities; Cardiovascular-cerebrovascular diseases; Real-world registry study; Disease-syndrome correlation
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Whole blood Whole blood Stool Lingual coating
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- T2DM-CVD, T2DM-CeVD，T2DM-CVD&CeVD: T2DM-CVD: Type 2 diabetes with ischemic cardiovascular disease (coronary artery disease/heart failure), excluding cerebrovascular involvement.
  2. T2DM-CeVD: Type 2 diabetes with ischemic cerebrovascular disease (ischemic stroke/TIA), excluding cardiovascular involvement.
  3. T2DM-CVD&CeVD: Type 2 diabetes comorbid with both ischemic cardiovascular and cerebrovascular diseases.

SUMMARY:
Explore the characteristics of TCM syndrome elements and distribution patterns of syndrome types in comorbid populations; Screen for "high-risk syndrome patterns" and frequently co-occurring complex syndromes; Identify characteristic syndrome patterns at key stages: acute phase, recovery phase, and upon occurrence of endpoint events; Investigate the temporal evolution of TCM syndrome patterns and the disease-syndrome correlation patterns in comorbid patients.

DETAILED DESCRIPTION:
A registry study of 12,000 real-world patients with comorbidities is conducted to collect and investigate the epidemiological characteristics of populations with "Tang-Nao" (diabetes with cerebrovascular disease), "Tang-Xin" (diabetes with cardiovascular disease), and triple comorbidities. Through syndrome epidemiology surveys, multi-timepoint cross-sectional investigations on the TCM syndrome of "Toxin Damaging Collaterals" are performed to explore the characteristics of TCM syndrome elements and distribution patterns of syndrome types in comorbid populations, screen "high-risk syndromes" and frequently co-occurring complex syndromes, identify characteristic syndromes at acute phase, recovery phase, and upon occurrence of endpoint events, and investigate the evolution of TCM syndromes and disease-syndrome correlation patterns in comorbid patients.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years Diagnosed with comorbidities relevant to "toxin-damaged collaterals" theory (e.g., type 2 diabetes mellitus with cardiovascular/cerebrovascular disease).

Voluntary participation with signed informed consent.

Exclusion Criteria:

* Acute infectious diseases, malignant tumors, or autoimmune disorders. Mental illness or cognitive impairment affecting symptom assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with comorbid chronic diseases (e.g., diabetes, coronary heart disease) who meet TCM "toxin-damaged collaterals" syndrome criteria.
Sampling Method: Non-Probability Sample
Enrollment: 12000 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2028-07-30 (Estimated); Study Completion 2028-07-30 (Estimated)

PRIMARY OUTCOMES:
Pattern (or Syndrome) Evolution Law in Traditional Chinese Medicine (TCM) | Baseline (enrollment, T0) and follow-up at 3 months (T1), 6 months (T2) with data collected through clinical visits and standardized syndrome assessment forms.
  Based on the TCM theory of "toxin-damaged collaterals," this outcome measures the dynamic changes in syndrome patterns (including qi deficiency, phlegm-dampness, heat-toxin, etc.) and their transition rules in patients with comorbidities. Assessment will use a standardized "Toxin-Damaged Collaterals Syndrome Collection Form", integrating four diagnostic methods (tongue coating, pulse, symptom scores, and syndrome differentiation results) at multiple follow-up time points to quantify syndrome evolution trends.